CLINICAL TRIAL: NCT03149575
Title: A Pivotal Randomized, Controlled Trial of VAL-083 in Patients With Recurrent Glioblastoma Who Have Failed Standard Temozolomide/Radiation Therapy and Bevacizumab (STAR-3)
Brief Title: VAL-083 Phase 3 Study in Temozolomide-Avastin (Bevacizumab) Recurrent GBM
Acronym: STAR-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Change in clinical development plan
Sponsor: DelMar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kintara Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DLM-16-002
Expanded Access: NCT03138629 (No longer available)
Record Dates: First submitted 2017-05-03; First posted 2017-05-11 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma Multiforme; Glioblastoma; Glioma; GBM; Brain Cancer
Keywords: Glioma; Glioblastoma; Glioblastoma multiforme; GBM; brain tumor; brain cancer; recurrent brain tumor; recurrent brain cancer; refractory brain tumor; refractory brain cancer; recurrent GBM; refractory GBM; recurrent glioma; refractory glioma; recurrent glioblastoma; refractory glioblastoma; recurrent glioblastoma multiforme; refractory glioblastoma multiforme; failed temodar; failed temozolomide; temodar refractory; temozolomide refractory; failed avastin; avastin refractory; failed bevacizumab; bevacizumab refractory; avastin failure; bevacizumab failure; STAR-3
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms | interventions — Dianhydrogalactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VAL-083, Dianhydrogalactitol (Experimental): Up to 120 eligible patients will be randomized to receive VAL-083.
  Interventions: Drug: VAL-083, Dianhydrogalactitol
- Physician's Choice of Salvage Therapy (Active Comparator): Up to 60 patients will be randomized to receive "Investigator's choice of salvage therapy" temozolomide, lomustine, or carboplatin
  Interventions: Drug: Physician's Choice of Salvage Therapy - temozolomide; Drug: Physician's Choice of Salvage Therapy - lomustine; Drug: Physician's Choice of Salvage Therapy - carboplatin

INTERVENTIONS:
Drug: VAL-083, Dianhydrogalactitol — VAL-083 given by intravenous infusion at a dose 40 mg/m2 IV on days 1, 2, and 3 of a 21-day treatment-cycle, for up to 12, 21-day treatment cycles
  Arms: VAL-083, Dianhydrogalactitol
Drug: Physician's Choice of Salvage Therapy - temozolomide — The product label for temozolomide (Temodar®) provides the following dosing information.
  Newly Diagnosed GBM: 75 mg/m2 for 42 days concomitant with focal radiotherapy followed by initial maintenance dose of 150 mg/m2 once daily for Days 1-5 of a 28-day cycle of Temodar® for 6 cycles.
  Refractory Anaplastic Astrocytoma: Initial dose 150 mg/m2 once daily for 5 consecutive days per 28-day treatment cycle.
  Arms: Physician's Choice of Salvage Therapy
Drug: Physician's Choice of Salvage Therapy - lomustine — The product label for lomustine (CeeNu; lomustine; CCNU) provides the following dosing information.
  The recommended dose of lomustine in adult and pediatric patients as a single agent in previously untreated patients is 130 mg/m2 as a single oral dose every 6 weeks In individuals with compromised bone marrow function, the dose should be reduced to 100 mg/m2 every 6 weeks.
  Arms: Physician's Choice of Salvage Therapy
Drug: Physician's Choice of Salvage Therapy - carboplatin — The product label for (Paraplatin) carboplatin Injection provides the following dosing information.
  As a single agent at a dosage of 360mg/m2 IV on day 1 every 28 days Alternatively, the carboplatin dose may be calculated by the Calvert formula below Calvert formula for carboplatin dosing: Total Dose (mg) = (target AUC) x (GFR + 25), where AUC = area under the curve and GFR = glomerular filtration rate.
  Arms: Physician's Choice of Salvage Therapy

SUMMARY:
This is an adaptive design, randomized controlled, Phase 3 clinical trial in patients with glioblastoma multiforme (GBM) or gliosarcoma (GS), previously treated with surgery (if appropriate), standard of care chemo-radiation with temozolomide, +/- adjuvant temozolomide, and bevacizumab and now has progressive disease during or after bevacizumab.

A total of up to 180 eligible patients with recurrent/progressive GBM or GS will be randomized to receive either the investigational drug (VAL-083) or "Investigator's choice of salvage therapy" as a contemporaneous control, in a 2:1 fashion. Up to 120 eligible patients will be randomized to receive VAL-083 at 40 mg/m2 IV on days 1, 2, and 3 of a 21-day treatment-cycle, for up to 12, 21-day treatment cycles or until they fulfill one of the criteria for study discontinuation. Up to 60 patients will be randomized to receive "Investigator's choice of salvage therapy", limited to temozolomide, lomustine, or carboplatin, until they fulfill one of the criteria for study discontinuation. The dose level for Investigator's choice salvage therapy (temozolomide, lomustine, or carboplatin), will be in accordance with the product label or institutional guidelines.

In both study arms, interval medical histories, targeted physical exams, neurologic evaluations, complete blood counts, and other laboratory and safety assessments will be performed approximately every 21-days while receiving treatment. Tumor assessments are to be performed approximately every 42 ± 7 days while remaining on study. The study is estimated to last approximately 20 months.

DETAILED DESCRIPTION:
This is an adaptive, randomized controlled, Phase 3 clinical trial in adult patients with histologically confirmed diagnosis of a recurrent glioblastoma multiforme (GBM) or gliosarcoma (GS), who have been previously treated with surgery (if appropriate), standard of care chemo-radiation with temozolomide, +/- adjuvant temozolomide, and bevacizumab and now have progressive disease during or after bevacizumab. Patients with prior low-grade glioma or anaplastic glioma are eligible, if histologic assessment demonstrates transformation to GBM or GS.

Treatment Groups: Eligible patients will be randomized to receive either the investigational drug (VAL-083) or "Investigator's choice of salvage therapy" as a contemporaneous control, in a 2:1 fashion. A total of up to 180 patients with recurrent/progressive GBM or GS will be enrolled; patients will be randomized to one of two treatment arms as follows:

Group 1: Up to 120 eligible patients will be randomized to receive VAL-083 at 40 mg/m2 IV on days 1, 2, and 3 of a 21-day treatment-cycle, for up to 12, 21-day treatment cycles or until they fulfill one of the criteria for study discontinuation (death, intolerable toxicities, investigator's judgment, or withdrawal of consent). In patients who demonstrate response, stable disease or who continue therapy at the discretion of the investigator following initial progression and tolerate therapy, permission to continue treatment beyond 12 cycles will be considered but will require consent of the Sponsor. VAL-083 will be administered as an IV infusion over 30-60 minutes.

Group 2: Up to 60 patients will be randomized to receive "Investigator's choice of salvage therapy" until they fulfill one of the criteria for study discontinuation (death, intolerable toxicities, investigator's judgment, or withdrawal of consent). "Investigator's choice of salvage therapy" will be limited to the following: temozolomide, lomustine, or carboplatin. The dose level for Investigator's choice salvage therapy (temozolomide, lomustine, or carboplatin), will be in accordance with the product label or institutional guidelines.

In both arms, disease status will be evaluated with clinical and imaging evaluation. Baseline total tumor burden must be assessed by MRI within 2 weeks prior to randomization. For patients randomized to VAL-083, post-baseline tumor assessments are to be performed prior to every other 21-day cycle for VAL-083, i.e., prior to Cycles 3, 5, etc., while the patient is receiving VAL-083 treatment, and then approximately every 42 ± 7 days while remaining on study. For patients randomized to the Physician's choice salvage therapy arm, post-baseline tumor assessments are to be performed approximately every 42 ± 7 days while remaining on study, as long as the patient continues to demonstrate response or stable disease or comes off the study.

In both study arms, assessments will include interval medical histories, Karnofsky Performance Status, physical and neurological examinations, vital signs, weight, adverse events, hematology and serum biochemistry, pregnancy test (females), urinalysis, chest x-ray and EKG approximately every 21-days while receiving treatment, as well as MDASI-BT self-reporting assessment when MRI tumor measurements are performed.

In a subgroup of 60 study subjects receiving VAL-083, blood samples will be obtained to determine population pharmacokinetics at pre-dose Cycle 1 Day 1, then at post-infusion on Cycle 1 Day 1, Cycle 1 Day 3, Cycle 2 Day 1 and Cycle 3 (or Cycle 4) Day 1 (or Day 3) in accordance with the study subject's assigned sampling block. EKGs will be taken pre-dose and approximately 10 minutes post-infusion Cycle 1 Day 1, prior to the 15 min (15 ± 5 min) blood draw for PK assessment, as well as pre-dose and approximately 10 minutes post-infusion Cycle 1 Day 3, prior to the 15 min (15 ± 5 min) blood draw for PK.

In a separate sub-group of 15 study subjects receiving VAL-083, blood will be drawn from Cycle 1 Day 1 and Cycle 1 Day 3 of dosing for determination of plasma levels of VAL-083 over the first 6 hours after the end of infusion (i.e., 0.25, 0.5, 1, 2, 4 and 6 hr). Trough levels 24 hr after infusion will also be obtained in these subjects. EKGs will be taken pre-dose and approximately 10 minutes post-infusion Cycle 1 Day 1, prior to the 15 min (15 ± 5 min) blood draw for PK assessment, as well as pre-dose and approximately 10 minutes post-infusion Cycle 1 Day 3, prior to the 15 min (15 ± 5 min) blood draw for PK.

Patients will be followed until death to ensure adequate power (90%) for the primary analysis.

Toxicity will be evaluated and documented using the NCI CTCAE version 4.

Quality of life will be evaluated using the MD Anderson Symptom Inventory-Brain Tumor (MDASI-BT). This questionnaire will be completed by patients at baseline and at the time of each imaging evaluation, until progression.

The study is estimated to take approximately 20 months, including 18 months to enroll 180 patients and another 2 months to reach 125 events (deaths).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must agree to testing of GBM tumor promoter methylation status of the MGMT gene and tumor (IDH1) gene mutation status. Tissue may be tested at study entry, if not done previously, or data may be obtained from last known test result for MGMT and IDH1. IDH1 status may be assessed at study entry, but MGMT status is required prior to randomization.
2. Agree to allow the sponsor to collect data on all GBM-related treatments received after the patient comes off the current study, and to collect survival data after the patient comes off the current study.
3. Patient must be ≥ 18 years old.
4. Histologically confirmed initial diagnosis of primary glioblastoma multiforme (GBM) or gliosarcoma (GS), now recurrent. Patients with recurrent/progressive disease whose initial diagnostic pathology confirmed GBM or GS will not need re-biopsy. Patients with prior low-grade glioma or anaplastic glioma are eligible, if histologic assessment demonstrates transformation to GBM or GS.
5. Patient has previously received standard of care chemo-radiation with temozolomide, ± adjuvant temozolomide and bevacizumab and now has radiographic evidence of recurrent/progressive GBM or GS during or after bevacizumab.
6. Patient must have bi dimensionally measurable disease, per the proposed Response Assessment in NeuroOncology (RANO; Appendix C) (Wen et al., 2010), with measurement of >1 cm in one diameter and ≤5 cm diameter in any plane on MRI performed within 2 weeks prior to randomization.
7. At least 4 weeks from last chemotherapy or bevacizumab (Avastin®) therapy (6 weeks for nitrosourea or mitomycin C), or for chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity, at least 2 weeks from last dose.
8. If the patient has been using the Optune™ device, it will be discontinued at least four days prior to commencing treatment with VAL-083, and the patient must have recovered from all treatment-related toxicities to Grade 1 or less.
9. Baseline MRI must be obtained ≥ 4 weeks after surgical resection but within 2 weeks prior to randomization.
10. Adequate recovery from all recent surgery is required; at least 1 week must have elapsed from the time of a minor surgery; at least 21 days must have elapsed from the time of a major surgery. Patients must have recovered from all surgery-related toxicities to Grade 1 or less.
11. Prior therapy with Laser-Induced Thermal Therapy (LITT) is allowed but at least 21 days must have elapsed from last LITT, with recovery from all LITT-related toxicities to Grade 1 or less and subsequent histologic documentation of recurrence.
12. Greater than 12 weeks from radiotherapy, to minimize the potential for MRI changes related to radiation necrosis that might be misdiagnosed as pseudoprogression of disease, unless the recurrence is a new lesion, outside the primary radiation field or the patient fulfills criteria for early progressive disease by RANO ((Wen et al., 2010); Appendix C).
13. Prior therapy with gamma knife or other focal high-dose radiation is allowed, but at least 2 weeks must have elapsed from the time of treatment, and the patient must have subsequent post-radiotherapy histologic documentation of recurrence in the irradiated field, unless the recurrence is a new lesion outside the irradiated field.
14. If receiving corticosteroids, patients must be on a stable or decreasing dose of corticosteroids for ≥ 5 days prior to baseline MRI.
15. At least 28 days or 5 half-lives (whichever is shorter) since prior investigational anti-cancer drugs. A minimum of 21 days between termination of the investigational drug and administration of VAL-083 is required.
16. Must have recovered from all treatment-related toxicities to Grade 1 or less.
17. Patients must have a Karnofsky performance status (KPS; Appendix D) of ≥ 70%
18. KPS must have been stable during the period from wash-out of prior therapy to randomization. A declining KPS is defined by reduction of 10 points or more over at least a 28-day period.
19. Patient must have a predicted life expectancy of at least 12 weeks.
20. Laboratory values as follows at screening and within 7 days of planned first dose of therapy:

    1. Absolute neutrophil count (ANC) ≥1500/μL.
    2. Hemoglobin (HgB) ≥9 g/dL.
    3. Platelets ≥100,000/μL (≥150,000/μL, if within 12 weeks of prior nitrosourea treatment).
    4. Serum creatinine ≤1.5 x upper limit of normal or creatinine clearance >60 mL/min (measured or calculated by the Cockcroft-Gault formula) (Cockcroft DW et al, 1976).
    5. AST, ALT must be <2 x ULN.
    6. Total bilirubin <1.5 x the institutional ULN, unless the subject has documented unconjugated bilirubin disorder such as Gilbert's syndrome.
    7. Subjects with known Gilbert's syndrome who have serum bilirubin ≤ 3 x ULN (NCI CTCAE v4.03 Grade 2) may be enrolled.
    8. International normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (aPTT) ≤ 1.5 x the ULN.
    9. QTc <450 msec on screening ECG.
21. No clinically significant cardiac conduction disorder on screening.
22. Female patients of child-bearing potential must have a negative serum or urine pregnancy test within 7 days prior to planned first dose of treatment, and agree to use dual method of contraception through 90 days after study drug treatment. Approved methods of contraception include an IUD with spermicide, a female condom with spermicide, a diaphragm with spermicide, a cervical cap with spermicide, use of a condom with spermicide by sexual partner or a sterile sexual partner. Women of childbearing potential are defined to include any female who:

    1. Has experienced menarche and has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy); and
    2. Is not post-menopausal (defined as amenorrhea >12 consecutive months).
23. If male, patient must be sterile or willing to use an approved method of contraception from the time of Informed Consent to 90 days after study drug treatment. Males must be willing to refrain from sperm donation within 90 days after study treatment.

Exclusion Criteria:

1. Current history of neoplasm other than the entry diagnosis. Exceptions are:

   1. Curatively treated basal cell/squamous cell skin cancer
   2. Carcinoma in situ of the cervix
   3. Patients with previous solid and hematologic tumors, that have been treated with no evidence of recurrence within the last 5 years, are permitted.
2. Evidence of diffuse subependymal disease or tumor in the brainstem, cerebellum, spinal cord, or CSF.
3. Radiological evidence of multifocal disease, tumors extending into or crossing the corpus callosum or leptomeningeal disease.
4. Need for urgent palliative intervention for primary disease (e.g., impending herniation).
5. Evidence of recent hemorrhage on baseline MRI of the brain with the following exceptions:

   1. Presence of hemosiderin.
   2. Resolving hemorrhagic changes related to surgery.
   3. Presence of punctate hemorrhage in the tumor.
6. Concurrent severe, intercurrent illness including, but not limited to unstable systemic disease, including ongoing or active infection, uncontrolled hypertension, serious cardiac arrhythmia requiring medication, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Any of the following cardiac conditions:

   1. History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, and/or stenting up to 12 weeks before Cycle 1, Day 1.
   2. Class III or IV heart failure as defined by the New York Heart Association functional classification system up to 6 months before Cycle 1, Day 1.
8. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair, or recent peripheral arterial thrombosis) within 6 months prior to Day 1 of treatment.
9. History of stroke or transient ischemic attack within 6 months prior to beginning treatment.
10. Patients receiving prohibited concomitant medications at the start of the study
11. Patients with steroid myopathy.
12. Patients who are HIV positive with an active AIDS-related illness are excluded; patients who are HIV positive but on stable therapy are not excluded.
13. Patients with a known sensitivity to any of the products to be administered during treatment and assessments.
14. Women who are pregnant or lactating.
15. Patients unable to undergo an MRI of the brain with contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Assessed approximately every 42 days for duration of study participation which is estimated to be 12 months
  Time from patient randomization to patient death

SECONDARY OUTCOMES:
Progression Free Survival | Assessed approximately every 42 days for duration of study participation which is estimated to be 12 months
  Time from patient randomization to first occurrence of disease progression (per RANO criteria) or death, whichever occurs first.
Duration of Response | Assessed approximately every 42 days for duration of study participation which is estimated to be 12 months
  Time from the patient's first occurrence of a documented, objective response (confirmed Complete Response or Partial Response) until the time of relapse (per RANO criteria) or death from any cause
Incidence of Treatment-Emergent Adverse Events (Overall Safety and Toxicity) | Assessed approximately every 42 days for duration of study participation which is estimated to be 12 months
  Time from patient randomization through 28 days following last study treatment received by patient. Safety will be assessed through summaries of AEs, changes in laboratory test results, ECGs, and changes in vital signs for all patients who receive any amount of VAL-083 or Physician's choice salvage therapy
Cmax | Assessed on Day 1 and Day 3 of Cycle 1 at pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration. Trough levels 24 hr after infusion on Day 1 will also be obtained in these subjects, prior to dosing on Day 2.
  Maximum observed plasma concentration of VAL-083 in a sub-group of 15 study subjects receiving VAL-083
Tmax | Assessed on Day 1 and Day 3 of Cycle 1 at pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration. Trough levels 24 hr after infusion on Day 1 will also be obtained in these subjects, prior to dosing on Day 2.
  Time of maximum observed plasma concentration of VAL-083 in a sub-group of 15 study subjects receiving VAL-083
AUClast | Assessed on Day 1 and Day 3 of Cycle 1 at pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration. Trough levels 24 hr after infusion on Day 1 will also be obtained in these subjects, prior to dosing on Day 2.
  Area under the concentration-time curve from pre-dose (time 0) to the time of the last quantifiable concentration of VAL-083 in plasma for a sub-group of 15 study subjects receiving VAL-083
AUCinf | Assessed on Day 1 and Day 3 of Cycle 1 at pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration. Trough levels 24 hr after infusion on Day 1 will also be obtained in these subjects, prior to dosing on Day 2.
  Area under the concentration-time curve extrapolated to infinity for VAL-083 in plasma of a sub-group of 15 study subjects receiving VAL-083
CL/F | Assessed on Day 1 and Day 3 of Cycle 1 at pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration. Trough levels 24 hr after infusion on Day 1 will also be obtained in these subjects, prior to dosing on Day 2.
  Total oral body clearance at steady state for VAL-083 in plasma of a sub-group of 15 study subjects receiving VAL-083
Mean Residence Time | Assessed on Day 1 and Day 3 of Cycle 1 at pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration. Trough levels 24 hr after infusion on Day 1 will also be obtained in these subjects, prior to dosing on Day 2.
  AUMC/AUC for VAL-083 in plasma of a sub-group of 15 study subjects receiving VAL-083, where AUMC is Area Under the Moment Curve
Vz | Assessed on Day 1 and Day 3 of Cycle 1 at pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration. Trough levels 24 hr after infusion on Day 1 will also be obtained in these subjects, prior to dosing on Day 2.
  Volume of distribution during the terminal phase of VAL-083 in plasma of a sub-group of 15 study subjects receiving VAL-083
Lambda z | Assessed on Day 1 and Day 3 of Cycle 1 at pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration. Trough levels 24 hr after infusion on Day 1 will also be obtained in these subjects, prior to dosing on Day 2.
  Terminal elimination rate constant determined by selection of at least 3 decreasing data points on the terminal phase of the concentration-time curve for VAL-083 in plasma of a sub-group of 15 study subjects receiving VAL-083
T 1/2 | Assessed on Day 1 and Day 3 of Cycle 1 at pre-dose, and 15, 30, 60, 120, 240 and 360 minutes after study drug administration. Trough levels 24 hr after infusion on Day 1 will also be obtained in these subjects, prior to dosing on Day 2.
  Terminal elimination half-life of VAL-083 in plasma of a sub-group of 15 study subjects receiving VAL-083
Quality of Life Assessment | Assessed approximately every 42 days for duration of study participation which is estimated to be 12 months
  Evaluate patient quality of life, using Quality of life will be evaluated using the MD Anderson Symptom Inventory-Brain Tumor (MDASI-BT), from time of patient randomization to first occurrence of disease progression (per RANO criteria) or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Butowski, M.D., Principal Investigator — University of California, San Francisco, California, USA 94143
Locations (5):
- United States (5):
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - University of California, San Francisco - Division of Neuro-Oncology, San Francisco, California
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Atlantic Neuroscience Institute - Brain Tumor Center of NJ, Summit, New Jersey
  - Dent Neurosciences Research Center, Amherst, New York

IPD SHARING:
Plan to Share IPD: No
The Clinical Study Report for this trial will be prepared upon completion of trial and provided to U.S. F.D.A. as required by applicable regulatory requirement(s). Each participating trial investigator will be provided a copy their patient data captured in the electronic data base for this trial. Data will include overall survival (OS), progression-free survival (PFS) at 6 months, median PFS, OS at 6 and 9 months, overall response rate (ORR), duration of response (DOR), disease control rate (DCR), occurrence of disease symptoms and evaluation of quality of life (QOL) measures during the progression-free period for VAL-083, compared to Investigator choice salvage therapy. Also, the safety and toxicity profile as well as pharmacokinetics of VAL-083 will be summarized.